CLINICAL TRIAL: NCT00401193
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study To Evaluate Efficacy and Safety of XP12B for the Treatment of Menorrhagia
Brief Title: Efficacy and Safety of XP12B in Women With Menorrhagia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XP12B-MR-301
Record Dates: First submitted 2006-11-09; First posted 2006-11-20 (Estimated); Results first posted 2010-02-24 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Menorrhagia; Heavy Menstrual Bleeding
Keywords: Menorrhagia; Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Tranexamic acid tablets
- 2 (Experimental)
  Interventions: Drug: Tranexamic acid tablets
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Tranexamic acid tablets — 3900 mg/Day
  Other Names: Lysteda; XP12B
  Arms: 1
Drug: Tranexamic acid tablets — 1950 mg/Day
  Other Names: Lysteda; XP12B
  Arms: 2
Drug: Placebo tablets
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether XP12B is effective and safe in the treatment of women with heavy menstrual bleeding associated with menorrhagia.

ELIGIBILITY:
Inclusion Criteria:

* Women with menorrhagia
* 18-49 years of age
* Regularly occurring menstrual periods

Exclusion Criteria:

* History or presence of clinically significant disease or abnormalities that may confound the study
* History of bilateral oophorectomy or hysterectomy
* Hormone therapy for birth control

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 304 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (79):
- United States (79):
  - Investigative Site, Birmingham, Alabama
  - Investigative Site, Phoenix, Arizona
  - Investigative Site, Tucson, Arizona
  - Investigative Site, Little Rock, Arkansas
  - Investigative Site, Searcy, Arkansas
  - Investigative Site, Los Alamitos, California
  - Investigative Site, Los Angeles, California
  - Investigative Site, San Diego, California
  - Investigative Site, Denver, Colorado
  - Investigative Site, Groton, Connecticut
  - Investigative Site, Gainesville, Florida
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Lighthouse PT, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Miami Beach, Florida
  - Investigative Site, New Port Richey, Florida
  - Investigative Site, Sarasota, Florida
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Decatur, Georgia
  - Investigative Site, Boise, Idaho
  - Investigative Site, Idaho Falls, Idaho
  - Investigative Site, Bloomington, Indiana
  - Investigative Site, Newton, Kansas
  - Investigative Site, Overland Park, Kansas
  - Investigative Site, Marrero, Louisiana
  - Investigative Site, Baltimore, Maryland
  - Investigative Site, Ann Arbor, Michigan
  - Investigative Site, Bingham Farms, Michigan
  - Investigative Site, Grand Rapids, Michigan
  - Investigative Site, Paw Paw, Michigan
  - Investigative Site, Saint Clair Shores, Michigan
  - Investigative Site, Kansas City, Missouri
  - Investigative Site, Missoula, Montana
  - Investigative Site, McCook, Nebraska
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, Lawrenceville, New Jersey
  - Investigative Site, Moorestown, New Jersey
  - Investigative Site, New Brunswick, New Jersey
  - Investigative Site, Albuquerque, New Mexico
  - Investigative Site, New York, New York
  - Investigative Site, Rochester, New York
  - Investigative Site, Durham, North Carolina
  - Investigative Site, Raleigh, North Carolina
  - Investigative Site, Winston-Salem, North Carolina
  - Investigative Site, Bismarck, North Dakota
  - Investigative Site, Cleveland, Ohio
  - Investigative Site, Gallipolis, Ohio
  - Investigative Site, Zanesville, Ohio
  - Investigative Site, Oklahoma City, Oklahoma
  - Investigative Site, Eugene, Oregon
  - Investigative Site, Portland, Oregon
  - Investigative Site, Levittown, Pennsylvania
  - Investigative Site, Philadelphia, Pennsylvania
  - Investigative Site, Phoenixville, Pennsylvania
  - Investigative Site, Strafford, Pennsylvania
  - Investigative Site, Wexford, Pennsylvania
  - Investigative Site, Wynnewood, Pennsylvania
  - Investigative Site, Greenville, South Carolina
  - Investigative Site, Sioux Falls, South Dakota
  - Investigative Site, Bristol, Tennessee
  - Investigative Site, Clarksville, Tennessee
  - Investigative Site, Nashville, Tennessee
  - Investigative Site, Austin, Texas
  - Investigative Site, Bryan, Texas
  - Investigative Site, Fort Worth, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, Plano, Texas
  - Investigative Site, Temple, Texas
  - Investigative Site, The Woodlands, Texas
  - Investigative Site, Waco, Texas
  - Investigative Site, Webster, Texas
  - Investigative Site, Pleasant Grove, Utah
  - Investigative Site, Salt Lake City, Utah
  - Investigative Site, West Jordan, Utah
  - Investigative Site, West Valley City, Utah
  - Investigative Site, Burlington, Vermont
  - Investigative Site, Norfolk, Virginia
  - Investigative Site, Richmond, Virginia
  - Investigative Site, Renton, Washington

REFERENCES:
- [Derived] Freeman EW, Lukes A, VanDrie D, Mabey RG, Gersten J, Adomako TL. A dose-response study of a novel, oral tranexamic formulation for heavy menstrual bleeding. Am J Obstet Gynecol. 2011 Oct;205(4):319.e1-7. doi: 10.1016/j.ajog.2011.05.015. Epub 2011 May 14. PMID 21777897
- [Derived] Lukes AS, Muse K, Richter HE, Moore KA, Patrick DL. Estimating a meaningful reduction in menstrual blood loss for women with heavy menstrual bleeding. Curr Med Res Opin. 2010 Nov;26(11):2673-8. doi: 10.1185/03007995.2010.526098. Epub 2010 Oct 13. PMID 20942615

RESULTS

PARTICIPANT FLOW:
Groups:
- 3900 mg/Day: Two 650 mg Lysteda (tranexamic acid) tablets taken 3 times daily (3900 mg/day) for a maximum of 5 days during monthly menstruation
- 1950 mg/Day: One 650 mg Lysteda (tranexamic acid) tablet and one matching placebo tablet taken 3 times daily (1950 mg/day) for a maximum of 5 days during monthly menstruation
- Placebo: Two placebo tablets taken 3 times daily for a maximum of 5 days during monthly menstruation
Period: Overall Study
Arm/Group | 3900 mg/Day | 1950 mg/Day | Placebo
Started | 118 | 117 | 69
Intent to Treat Population | 115 | 115 | 67
Modified Intent to Treat Population | 112 | 115 | 67
Completed | 103 | 106 | 63
Not Completed | 15 | 11 | 6
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — Lost to Follow-up | 6 | 5 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Other Event | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3900 mg/Day | 1950 mg/Day | Placebo | Total
Number analyzed (Participants) | 115 | 115 | 67 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] — Intent to Treat Population
  years | 39 (6) | 40 (6) | 39 (6) | 39 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 115 | 67 | 297
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction From Baseline in Menstrual Blood Loss (MBL)
Description: reduction of menstrual blood loss in mL
Time Frame: Baseline MBL over 3 menstrual cycles
Population: modified intent to treat population
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | 3900 mg/Day | 1950 mg/Day | Placebo
Number analyzed (Participants) | 112 | 115 | 67
mL | 65 (51) | 44 (57) | 7 (46)

2. Secondary Outcome: Patient Reported Outcome Measure of Limitations in Social or Leisure Activities Associated With Heavy Menstrual Bleeding
Description: A positive unit change of the mean relects an improvement from baseline. Patient reported outcome scores had the following response categories: 1=not limited at all; 2=slightly limited; 3=moderately limited; 4=quite a bit limited; and 5=extremely limited
Time Frame: Baseline scores over 3 menstrual cycles
Population: modified intent to treat population (reflects those subjects who met the criteria for the primary efficacy analysis)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3900 mg/Day | Placebo
Number analyzed (Participants) | 112 | 66
units on a scale | 1.0 (1.1) | 0.4 (0.8)

3. Secondary Outcome: Patient Reported Outome Measure of Limitations in Physical Activities Associated With Heavy Menstrual Bleeding
Description: as for outcome 2
Time Frame: Baseline scores over 3 menstrual cycles
Population: modified intent to treat population (reflects those subjects who met the criteria for the primary efficacy analysis)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3900 mg/Day | Placebo
Number analyzed (Participants) | 112 | 66
units on a scale | 0.9 (1.0) | 0.3 (0.8)

4. Secondary Outcome: Responder Analysis - Reduction in Large Stains
Description: Percentage of subjects who experienced a reduction from baseline in the frequency of large stains
Time Frame: Baseline over 3 mentrual cycles
Population: modified intent to treat population (reflects those subjects who met the criteria for the primary efficacy analysis)
Measure: Number; unit: percentage of participants
Arm/Group | 3900 mg/Day | Placebo
Number analyzed (Participants) | 111 | 67
percentage of participants | 64 | 52

ADVERSE EVENTS:
Arm/Group | 3900 mg/Day | 1950 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/115 | 1/115 | 0/67
Other Adverse Events (participants affected / at risk) | 97/115 | 104/115 | 56/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3900 mg/Day (N=115) | 1950 mg/Day (N=115) | Placebo (N=67)
Chest Pain (General disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Ovarian Torsion (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3900 mg/Day (N=115) | 1950 mg/Day (N=115) | Placebo (N=67)
Abdominal Pain (Gastrointestinal disorders) | 23 | 24 | 15
Anemia (Blood and lymphatic system disorders) | 1 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 20 | 20 | 7
Fatigue (General disorders) | 4 | 13 | 3
Headache (Nervous system disorders) | 48 | 54 | 26
Migraine (Nervous system disorders) | 7 | 7 | 4
Muscle Cramps & Spasms (Musculoskeletal and connective tissue disorders) | 6 | 3 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 | 15 | 2
Nasal & Sinus Symptoms (Immune system disorders) | 16 | 35 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other